CLINICAL TRIAL: NCT00116623
Title: Magnesium Sulfate Versus Indomethacin for Preterm Labor
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding completed
Sponsor: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 704914
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Labor, Premature
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Indomethacin; Magnesium Sulfate

INTERVENTIONS:
Drug: Indomethacin
Drug: Magnesium sulfate

SUMMARY:
The purpose of this study is to investigate the efficacy of Indomethacin compared to Magnesium Sulfate (MgSO4) in reducing neonatal morbidity through a prospective double blind randomized clinical trial. The specific aim of the project is to test the hypothesis that Indomethacin, compared to MgSO4, will decrease the proportion of neonates diagnosed with major complications or death.

ELIGIBILITY:
Inclusion Criteria:

* Initial episode of preterm labor for enrollment
* The diagnosis of preterm labor
* Gestational age between 24 and 32 weeks
* Singleton or twin gestation
* The ability to understand the requirements of the study

Exclusion Criteria:

* Cervical dilation >5 cms
* Suspected chorioamnionitis
* Fetal distress
* Vaginal bleeding
* Severe pre-eclampsia
* History of gastrointestinal bleeding
* Abnormal renal function
* Suspicion of fetal malformation by ultrasound
* Known allergy to, or intolerance of, Magnesium sulfate and/or Indomethacin
* Documented rupture of amniotic membranes
* Multiple gestations of triplets or more.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-02; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George A Macones, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046